CLINICAL TRIAL: NCT07111871
Title: Understanding Care Pathways for Older People on Anticoagulant or Antiplatelet Medications With Falls and Head Injury
Brief Title: Healthcare Services for Older People Who Have Fallen With Potential Head Injury
Acronym: Anti-HI-Falls
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHU/2025/35
Record Dates: First submitted 2025-07-14; First posted 2025-08-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Older Adults (65 Years and Older); Falls; Head Injury
Keywords: Older People; Anticoagulants; Antiplatelets; Falls; Head injury; Care pathways
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NHS Healthcare workers: NHS health professionals working in any sectors (primary, secondary, tertiary) within Hampshire and Isle of Wight that assess older people (age >65 who have had a fall as part of their job role

SUMMARY:
Every year, one in three older people (>65 years old) experience a fall. Older people may have long-term health conditions and take medications that can increase their risk of bleeding (blood thinners). The UK national guidelines recommend that older people who are on blood thinning medications should have a CT head scan considered due to concerns of a brain bleed if they have hit their head after a fall. Many older people are therefore brought into hospital for assessment. However, the risk of bleeding in the brain is very low especially if older people do not have any symptoms such as loss of consciousness, weakness, headaches or vomiting. Some people could experience long waits in the emergency department or end up being admitted to hospital unnecessarily. This could worsen mobility, cause confusion, pressure sores or infections in older people.

More importantly, older people should have a comprehensive falls assessment to reduce their risk of future falls and have their medications reviewed after experiencing a fall. These assessments could potentially take place in their own homes if they prefer, rather than in hospital. Yet, current healthcare services outside the hospital setting may not be set up to manage an older person after fall.

Using an online survey, the investigators want to understand how current healthcare services in the Hampshire and Isle of Wight (HIOW) region work to look after older people who have had a fall. The study will focus particularly on older people taking blood thinning medications who may have a head injury but do not have any symptoms. The investigators will ask NHS workers what their role is, where they work and what they do when assessing an older person who has fallen if there is a concern about head injury. The survey will also ask participants to describe what challenges they may face, and if they have any suggestions to improve the care for older people.

This study will help the investigators understand what services are available in our current healthcare system for older people on blood thinning medications who have fallen and may have a head injury. The investigators hope that the results will help improve how healthcare services can work together with older people and their closed ones to provide care based on what matters most to them in their preferred place of care. This could reduce unnecessary use of emergency services and hospital admissions for older people.

DETAILED DESCRIPTION:
Falls is a common problem that impact older people (>65 years old). One in three people over the age of 65, and approximately half of those aged 80 and above experience a fall each year. Falls can have devastating consequences and lead to head injury, bone fractures, loss of confidences and death. Up to a third of older people who fall are taking anticoagulant and/or antiplatelet medications (blood thinners) for manage long-term conditions such as atrial fibrillation, ischaemic heart disease, and stroke. Due to concerns of bleeding in the brain after a fall, current national guidelines recommend that older people on anticoagulant or antiplatelet medications should be taken to hospital for assessment to consider whether CT head scan is needed. This is recommended even if patients do not have any signs of head injury, or worrying symptoms such as headache, weakness, or vomiting.

Performing a CT head on every older person on blood thinners who has fallen is not cost-effective nor practical. Current evidence suggests that the risk of bleeding in the brain is low (approximately 5%) in older people. Studies have reported that there is no increased risk of bleeding in the brain even if older people are on blood thinners, particularly if they do not have any worrying symptoms. However, many older people are often brought into hospital despite having no symptoms of head injury. This can lead to long waiting times to be seen in the Emergency Department.

For some older people, unnecessary hospital admissions can have a negative impact on their ability to walk, cause infections, confusions and pressure sores. The risk of being in hospital may not outweigh the small risk of having a brain bleed, particularly if they do not have any signs of head injury or worrying symptoms. Older people could have a comprehensive falls assessment, review of medications and follow-up outside of the hospital setting.

Alternative services to hospital admission for older people have been developed in the recent years to support people in their preferred place, and reduce pressures in the emergency departments. We know from clinical practice that services such as urgent community response teams, acute frailty wards, same day emergency care or hospital at homes often manage older people who have had a fall with possible head injury. Yet, no research studies have specifically reviewed care pathways and outcomes for older people on anticoagulant or antiplatelet medications who have had a fall and head injury with no symptoms outside the hospital.

We want to understand how the services in Hampshire and Isle of Wight region are working to support older people on anticoagulant and antiplatelet medications who have had a fall with head injury. We want to know what challenges healthcare workers experience, and what suggestions they have to improve this. This can help us improve service delivery for older people.

ELIGIBILITY:
Inclusion Criteria:

* • Aged 18 years or above

  * Healthcare professional whose primary employment is within HIOW
  * Have experience reviewing older adults on anticoagulant or antiplatelet medications who have had a fall as part of their job role
  * Confirmed consent to participate on the completed survey

Exclusion Criteria:

* • Did not consent to participate on the completed survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a cross-sectional mixed-methods online survey involving NHS healthcare professionals working in HIOW ICS across all relevant sectors. This could include those working in (but not limited to):
  * Acute hospitals including ED, Acute Medical Unit, Older Persons/Geriatric departments, Same Day Emergency Care services
  * Primary care services including out of hours
  * Community health services (urgent community response services, acute frailty wards, hospital at home, urgent treatment centres)
  * South Central Ambulance Services (SCAS) and 111 emergency services
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Current healthcare service pathways | 24 months
  Describe healthcare services and clinical pathways across primary care, community care and secondary care services for older people following fall. This will include frequency and proportions of healthcare professionals' roles, experience, and assessment of an older person on anticoagulant or antiplatelet medications following a fall with asymptomatic head injury including availability of falls assessment and medication reviews.

SECONDARY OUTCOMES:
Challenges or barriers experienced by healthcare professionals | 24 months
  Understand experiences faced by healthcare professionals through qualitative analysis of open-ended questions

CONTACTS AND LOCATIONS:
Overall Officials: Qian Yue Tan, PhD BM, Study Chair — Portsmouth Hospitals University NHS Trust
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be anonymised and will not be shared outside the research team.